CLINICAL TRIAL: NCT00363415
Title: A Randomized Phase 3 Trial of Alimta (Pemetrexed) and Carboplatin Versus Etoposide and Carboplatin in Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of Pemetrexed and Carboplatin Compared With Etoposide Carboplatin to Treat Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9691; H3E-MC-JMHO
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2009-10-06 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Pemetrexed; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: pemetrexed; Drug: carboplatin
- B (Active Comparator)
  Interventions: Drug: etoposide; Drug: carboplatin

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 6 cycles
  Other Names: LY231514; Alimta
  Arms: A
Drug: etoposide — 100 mg/m2, intravenous (IV), days 1-3 x 6 cycles
  Arms: B
Drug: carboplatin — Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles

SUMMARY:
This study is a Phase 3, global, multi-center, open-label study of patients with extensive-stage small cell lung cancer. Eligible patients will be randomly assigned to receive either pemetrexed plus carboplatin or etoposide plus carboplatin. It is anticipated that pemetrexed plus carboplatin will offer similar survival benefits as compared to etoposide plus carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of extensive stage small cell lung cancer (SCLC)
* Capable of self-care but may be unable to carry out any work activities.
* No prior anticancer therapy for SCLC

Exclusion Criteria:

* have previously participated in a study involving pemetrexed
* have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (189):
- United States (54):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poway, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scarborough, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sparta, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zanesville, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Stroudsburg, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ephrata, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilkes-Barre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bahía Blanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucumain
- Australia (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coffs Harbour, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Macquarie, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brisbane, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chermisdie, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redcliffe, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Brisbane, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Townsville, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodville, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hobart, Tasmania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wodonga, Victoria
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florianópolis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaú
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clichy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
- Germany (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Borstel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gauting
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Regensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stralsund
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marousi Attikis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pylaia/Thessaloniki
- Hungary (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deszk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szombathely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Törökbálint
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- India (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludhiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monteforte Irpino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ravenna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sisto
- Netherlands (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harderwijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heerlen
- New Zealand (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow-Nowa Huta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otwock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin-Zdunowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zabrze-Biskupice
- Portugal (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria da Feira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vila Nova de Gaia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Engel's
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murmansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parktown
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barakaldo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaragoza
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besevler/Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samsun
- United Kingdom (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Truro, Cornwall
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelmsford, Essex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

REFERENCES:
- [Derived] Ventz S, Khozin S, Louv B, Sands J, Wen PY, Rahman R, Comment L, Alexander BM, Trippa L. The design and evaluation of hybrid controlled trials that leverage external data and randomization. Nat Commun. 2022 Oct 2;13(1):5783. doi: 10.1038/s41467-022-33192-1. PMID 36184621
- [Derived] Socinski MA, Smit EF, Lorigan P, Konduri K, Reck M, Szczesna A, Blakely J, Serwatowski P, Karaseva NA, Ciuleanu T, Jassem J, Dediu M, Hong S, Visseren-Grul C, Hanauske AR, Obasaju CK, Guba SC, Thatcher N. Phase III study of pemetrexed plus carboplatin compared with etoposide plus carboplatin in chemotherapy-naive patients with extensive-stage small-cell lung cancer. J Clin Oncol. 2009 Oct 1;27(28):4787-92. doi: 10.1200/JCO.2009.23.1548. Epub 2009 Aug 31. PMID 19720897
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received at least one dose of study drug were, per protocol, the patient population used for the summary of safety data (eg, Serious Adverse Events).
Groups:
- Pemetrexed + Carboplatin: Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles Carboplatin: Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles
- Etoposide + Carboplatin: Etoposide: 100 mg/m2, intravenous (IV), days 1-3 x 6 cycles Carboplatin: Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Started | 453 | 455
Received at Least One Dose of Study Drug | 433 | 447
Completed | 92 | 206
Not Completed | 361 | 249
Not completed — Progressive Disease | 196 | 107
Not completed — Sponsor Decision | 67 | 31
Not completed — Death | 32 | 29
Not completed — Adverse Event | 24 | 15
Not completed — Physician Decision | 18 | 35
Not completed — Entry Criteria Not Met | 11 | 10
Not completed — Withdrawal by Subject | 9 | 15
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin | Total
Number analyzed (Participants) | 453 | 455 | 908
Age, Customized [Number; unit: participants]
  <=65 years | 267 | 275 | 542
  >65 years | 186 | 180 | 366
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 125 | 253
  Male | 325 | 330 | 655
Region of Enrollment [Number; unit: participants]
  United States | 92 | 83 | 175
  Portugal | 9 | 7 | 16
  Taiwan | 11 | 12 | 23
  Greece | 7 | 8 | 15
  Spain | 16 | 21 | 37
  Russian Federation | 30 | 16 | 46
  Italy | 7 | 8 | 15
  India | 12 | 14 | 26
  France | 19 | 10 | 29
  Australia | 21 | 19 | 40
  South Africa | 0 | 1 | 1
  Netherlands | 17 | 17 | 34
  China | 14 | 18 | 32
  Korea, Republic of | 17 | 15 | 32
  Turkey | 15 | 13 | 28
  Austria | 5 | 14 | 19
  United Kingdom | 16 | 18 | 34
  Hungary | 19 | 13 | 32
  Argentina | 2 | 6 | 8
  Belgium | 12 | 17 | 29
  Brazil | 4 | 7 | 11
  Poland | 29 | 34 | 63
  Romania | 20 | 23 | 43
  Germany | 58 | 59 | 117
  New Zealand | 1 | 2 | 3
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 133 | 121 | 254
    1 - Ambulatory, Restricted Strenuous Activity | 265 | 277 | 542
    2 - Ambulatory, No Work Activities | 54 | 55 | 109
    3 - Partially Confined to Bed, Limited Self Care | 1 | 0 | 1
    Not Reported | 0 | 2 | 2
History of Brain Metastases [Number; unit: participants]
  No | 410 | 412 | 822
  Yes | 43 | 41 | 84
  Not Reported | 0 | 2 | 2
Race/Ethnicity [Number; unit: participants]
  Caucasian | 391 | 379 | 770
  East Asian | 43 | 49 | 92
  West Asian | 12 | 12 | 24
  African | 5 | 8 | 13
  Hispanic | 1 | 5 | 6
  Aboriginal and/or Torres Strait Islander | 0 | 2 | 2
  Native American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 19.6 months)
Population: Number of participants with events. In the pemetrexed+carboplatin group, 242 participants were censored. In the etoposide+carboplatin group, 288 participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 211 | 167
months | 8.1 [7.3 to 9.1] | 10.6 [9.7 to 11.6]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.01, Log Rank; Hazard Ratio (HR) = 1.56, 95% CI [1.27 to 1.92]

2. Secondary Outcome: Overall Survival (Subgroups)
Description: The effects of individual baseline factors (sex, race, Eastern Cooperative Oncology Group (ECOG) performance, region, lactate dehydrogenase (LDH), age, number of metastatic sites, and history of brain metastases) on overall survival are reported. For two subgroups - LDH<=upper limit of normal and brain metastases=yes, the upper limits of the 95% confidence interval were not calculable for the etoposide+carboplatin group - instead the number of participants in these two subgroups are presented as a post-hoc outcome measure.
Time Frame: baseline to date of death from any cause (up to 19.6 months)
Population: Number of randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 453 | 455
months
  Sex: Male (n=325, n=330) | 8.2 [7.2 to 9.1] | 10.4 [9.3 to 11.5]
  Sex: Female (n=128, n=125) | 8.1 [7.2 to 9.7] | 11.6 [10.3 to 13.0]
  Race: Caucasian (n=391, n=379) | 8.2 [7.6 to 9.4] | 11.2 [9.9 to 12.0]
  Race: Non-Caucasian (n=62, n=76) | 7.1 [5.7 to 9.1] | 8.7 [7.2 to 14.9]
  ECOG: 0 or 1 (n=398, n=398) | 8.5 [7.8 to 9.4] | 11.3 [10.1 to 12.0]
  ECOG: 2 (n=54, n=55) | 6.2 [3.7 to 7.3] | 5.2 [3.9 to 9.5]
  Region: United States (n=92, n=83) | 8.1 [7.3 to 9.8] | 11.3 [9.3 to 12.9]
  Region: European Union (n=279, n=278) | 8.5 [7.2 to 9.7] | 11.2 [9.5 to 12.9]
  Region: Intercontinential Region (n=82, n=94) | 7.2 [6.1 to 8.6] | 9.9 [8.5 to 11.9]
  LDH: >Upper Limit of Normal (n=276, n=273) | 7.2 [6.5 to 8.3] | 9.3 [8.0 to 10.4]
  Age: <= 65 years (n=267, n=275) | 8.4 [7.5 to 9.7] | 11.5 [10.3 to 12.9]
  Age: >65 years (n=186, n=180) | 7.7 [7.1 to 9.0] | 9.7 [8.7 to 11.3]
  Number Metastatic Sites: <=2 (n=172, n=204) | 10.0 [8.6 to 13.5] | 11.5 [10.1 to 13.2]
  Number Metastatic Sites: >=3 (n=273, n=246) | 7.7 [7.2 to 8.2] | 10.3 [9.3 to 11.3]
  History of Brain Metastases: No (n=410, n=412) | 8.2 [7.3 to 9.1] | 10.6 [9.5 to 11.6]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for Sex: Male
Statistical Analysis 2: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.023, Log Rank — P-value for Sex: Female
Statistical Analysis 3: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for Race: Caucasian
Statistical Analysis 4: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.030, Log Rank — P-value for Race: Non-Caucasian
Statistical Analysis 5: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for ECOG (Eastern Cooperative Oncology Group) Performance Status: 0 or 1
Statistical Analysis 6: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.519, Log Rank — P-value for ECOG (Eastern Cooperative Oncology Group) Performance Status: 2
Statistical Analysis 7: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.084, Log Rank — P-value for Region: United States
Statistical Analysis 8: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.001, Log Rank — P-value for Region: European Union
Statistical Analysis 9: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.003, Log Rank — P-value for Region: Intercontinental Region
Statistical Analysis 10: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.005, Log Rank — P-value for LDH (lactate dehydrogenase): >Upper Limit of Normal
Statistical Analysis 11: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for Age: <=65 years
Statistical Analysis 12: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.013, Log Rank — P-value for Age: >65 years
Statistical Analysis 13: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p = 0.092, Log Rank — P-value for Number Metastatic Sites: <=2
Statistical Analysis 14: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for Number Metastatic Sites: >=3
Statistical Analysis 15: Comparison: Pemetrexed + Carboplatin vs Etoposide + Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — P-value for History of Brain Metastases: No

3. Secondary Outcome: Progression Free Survival
Description: The period from study entry until disease progression, death or date of last contact.
Time Frame: baseline to measured progressive disease (up to 14.7 months)
Population: All randomized participants. Number of participants censored: 113 in Pemetrexed+Carboplatin; 150 in Etoposide+Carboplatin.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 453 | 455
months | 3.8 [3.5 to 4.2] | 5.4 [5.2 to 5.7]

4. Secondary Outcome: Change From Baseline to Each Cycle in Functional Assessment of Cancer Therapy - Lung (FACT-L)
Description: FACT-L measures following domains of health-related quality of life (HR-QL): physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns of lung cancer. Total scores range from 0 to 136, with higher scores representing better HR-QL. A clinically meaningful change is considered to be 5 points.
Time Frame: baseline and 6 cycles (21-day cycles)
Population: Number of randomized participants with baseline and non-missing value at respective cycle.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 384 | 383
units on a scale
  Baseline (n=384, n=383) | 87.42 (15.40) | 87.79 (16.63)
  Cycle 1 Change from Baseline (n=270, n=275) | -0.22 (12.48) | 1.55 (11.11)
  Cycle 2 Change from Baseline (n=283, n=310) | 0.17 (13.72) | 1.73 (12.73)
  Cycle 3 Change from Baseline (n=225, n=277) | 0.06 (14.61) | 1.70 (13.98)
  Cycle 4 Change from Baseline (n=199, n=259) | -0.14 (15.28) | 1.69 (13.42)
  Cycle 5 Change from Baseline (n=140, n=203) | 0.27 (16.34) | 1.94 (14.06)
  Cycle 6 Change from Baseline (n=98, n=146) | 0.34 (17.56) | 3.73 (14.97)

5. Secondary Outcome: Overall Survival (Subgroups: LDH<=Upper Limit of Normal and History of Brain Metastases=Yes)
Description: The effects of individual baseline factors (lactate dehydrogenase (LDH) and history of brain metastases) on overall survival are reported. The Upper Limits of the 95% Confidence Intervals were not calculable for these factors in the Etoposide+Carboplatin group. The number of participants in these subgroup are instead presented as a Post-Hoc Outcome Measure.
Time Frame: baseline to date of death due to any cause (up to 19.6 months)
Population: The upper limit of the 95% Confidence Intervals (CI) were not calculable for these two subgroups in the etoposide+carboplatin group so medians and lower limits of the 95% CI are not presented. A post-hoc outcome measure table provides the number of participants in each subgroup.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 0 | 0

6. Post Hoc Outcome: Number of Participants in Subgroups: LDH<=Upper Limit of Normal and History of Brain Metastases=Yes
Description: Number of participants with Low Density Lipoprotein <=upper limit of normal and the number of participants with a history of brain metastases. This post-hoc outcome replaces the one for Overall Survival (Subgroups: LDH<=Upper Limit of Normal and History of Brain Metastases=Yes).
Time Frame: baseline to date of death due to any cause (up to 19.6 months)
Population: Number of randomized participants.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Number analyzed (Participants) | 453 | 455
participants
  LDH: <=Upper Limit of Normal | 167 | 169
  History of Brain Metastases: Yes | 43 | 41

ADVERSE EVENTS:
Groups:
- Pemetrexed + Carboplatin: Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles Carboplatin: Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles (Participants who received at least one dose of study drug)
- Etoposide + Carboplatin: Etoposide: 100 mg/m2, intravenous (IV), days 1-3 x 6 cycles Carboplatin: Area under the curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles.
  (Participants who received at least one dose of study drug)
Arm/Group | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Serious Adverse Events (participants affected / at risk) | 150 | 134
Other Adverse Events (participants affected / at risk) | 425 | 438
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Agranulocytosis (Blood and lymphatic system disorders) | 0/433 (0) | 1/447 (1)
Anaemia (Blood and lymphatic system disorders) | 18/433 (20) | 7/447 (7)
Bone marrow failure (Blood and lymphatic system disorders) | 1/433 (1) | 0/447 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7/433 (8) | 14/447 (14)
Leukopenia (Blood and lymphatic system disorders) | 4/433 (4) | 4/447 (4)
Neutropenia (Blood and lymphatic system disorders) | 11/433 (12) | 19/447 (21)
Splenic infarction (Blood and lymphatic system disorders) | 2/433 (2) | 0/447 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 15/433 (18) | 7/447 (8)
Acute coronary syndrome (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Acute left ventricular failure (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Acute myocardial infarction (Cardiac disorders) | 1/433 (1) | 1/447 (1)
Angina pectoris (Cardiac disorders) | 1/433 (1) | 1/447 (1)
Angina unstable (Cardiac disorders) | 0/433 (0) | 2/447 (2)
Atrial fibrillation (Cardiac disorders) | 5/433 (5) | 0/447 (0)
Atrial flutter (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Cardiac arrest (Cardiac disorders) | 2/433 (2) | 1/447 (1)
Cardiac failure (Cardiac disorders) | 2/433 (2) | 0/447 (0)
Cardiac failure acute (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Cardiac failure congestive (Cardiac disorders) | 1/433 (1) | 1/447 (1)
Cardiac fibrillation (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2/433 (2) | 1/447 (1)
Coronary artery insufficiency (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Left ventricular dysfunction (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Myocardial infarction (Cardiac disorders) | 4/433 (4) | 1/447 (1)
Myocardial ischaemia (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Supraventricular tachycardia (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Ventricular fibrillation (Cardiac disorders) | 1/433 (1) | 0/447 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1/433 (1) | 0/447 (0)
Vertigo (Ear and labyrinth disorders) | 1/433 (1) | 0/447 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1/433 (1) | 2/447 (2)
Eyelid ptosis (Eye disorders) | 0/433 (0) | 1/447 (1)
Retinal detachment (Eye disorders) | 1/433 (1) | 0/447 (0)
Abdominal pain (Gastrointestinal disorders) | 4/433 (4) | 1/447 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2/433 (2) | 2/447 (2)
Colitis (Gastrointestinal disorders) | 2/433 (2) | 0/447 (0)
Constipation (Gastrointestinal disorders) | 4/433 (4) | 4/447 (4)
Diarrhoea (Gastrointestinal disorders) | 11/433 (11) | 3/447 (3)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0/433 (0) | 1/447 (1)
Dysphagia (Gastrointestinal disorders) | 3/433 (3) | 1/447 (1)
Gastric ulcer (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Gastritis (Gastrointestinal disorders) | 0/433 (0) | 1/447 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Nausea (Gastrointestinal disorders) | 15/433 (18) | 2/447 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 0/433 (0) | 2/447 (2)
Oral discomfort (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0/433 (0) | 2/447 (2)
Proctitis (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1/433 (1) | 0/447 (0)
Vomiting (Gastrointestinal disorders) | 11/433 (11) | 4/447 (4)
Asthenia (General disorders) | 4/433 (4) | 2/447 (2)
Chest discomfort (General disorders) | 0/433 (0) | 1/447 (1)
Chest pain (General disorders) | 4/433 (4) | 4/447 (4)
Condition aggravated (General disorders) | 0/433 (0) | 1/447 (1)
Fatigue (General disorders) | 3/433 (3) | 2/447 (2)
General physical health deterioration (General disorders) | 1/433 (1) | 0/447 (0)
Malaise (General disorders) | 2/433 (2) | 0/447 (0)
Mucosal inflammation (General disorders) | 0/433 (0) | 1/447 (1)
Pain (General disorders) | 1/433 (1) | 0/447 (0)
Performance status decreased (General disorders) | 0/433 (0) | 2/447 (2)
Pyrexia (General disorders) | 3/433 (3) | 5/447 (6)
Sudden death (General disorders) | 0/433 (0) | 1/447 (1)
Visceral oedema (General disorders) | 0/433 (0) | 1/447 (1)
Hepatic failure (Hepatobiliary disorders) | 0/433 (0) | 1/447 (1)
Hepatic pain (Hepatobiliary disorders) | 1/433 (1) | 0/447 (0)
Anaphylactic shock (Immune system disorders) | 1/433 (1) | 0/447 (0)
Drug hypersensitivity (Immune system disorders) | 0/433 (0) | 1/447 (1)
Hypersensitivity (Immune system disorders) | 0/433 (0) | 1/447 (1)
Bacterial sepsis (Infections and infestations) | 0/433 (0) | 1/447 (1)
Bronchopneumonia (Infections and infestations) | 1/433 (1) | 1/447 (1)
Candidiasis (Infections and infestations) | 0/433 (0) | 1/447 (1)
Catheter related infection (Infections and infestations) | 1/433 (1) | 0/447 (0)
Cellulitis (Infections and infestations) | 0/433 (0) | 1/447 (1)
Device related infection (Infections and infestations) | 0/433 (0) | 1/447 (1)
Diverticulitis (Infections and infestations) | 1/433 (1) | 1/447 (1)
Empyema (Infections and infestations) | 3/433 (3) | 2/447 (3)
Encephalitis herpes (Infections and infestations) | 0/433 (0) | 1/447 (1)
Enteritis infectious (Infections and infestations) | 1/433 (1) | 0/447 (0)
Febrile infection (Infections and infestations) | 0/433 (0) | 1/447 (1)
Gastroenteritis (Infections and infestations) | 1/433 (1) | 0/447 (0)
Herpes zoster (Infections and infestations) | 0/433 (0) | 1/447 (1)
Infection (Infections and infestations) | 1/433 (1) | 0/447 (0)
Klebsiella sepsis (Infections and infestations) | 1/433 (1) | 0/447 (0)
Lower respiratory tract infection (Infections and infestations) | 2/433 (2) | 0/447 (0)
Lung abscess (Infections and infestations) | 0/433 (0) | 1/447 (1)
Lung infection (Infections and infestations) | 2/433 (2) | 0/447 (0)
Necrotising fasciitis (Infections and infestations) | 1/433 (1) | 0/447 (0)
Neutropenic sepsis (Infections and infestations) | 1/433 (1) | 2/447 (2)
Pneumonia (Infections and infestations) | 20/433 (24) | 15/447 (16)
Pneumonia necrotising (Infections and infestations) | 0/433 (0) | 1/447 (1)
Pneumonia primary atypical (Infections and infestations) | 1/433 (1) | 1/447 (1)
Pneumonia staphylococcal (Infections and infestations) | 0/433 (0) | 1/447 (1)
Pseudomembranous colitis (Infections and infestations) | 1/433 (1) | 0/447 (0)
Respiratory tract infection (Infections and infestations) | 1/433 (1) | 3/447 (3)
Sepsis (Infections and infestations) | 5/433 (5) | 5/447 (5)
Septic shock (Infections and infestations) | 3/433 (3) | 0/447 (0)
Staphylococcal infection (Infections and infestations) | 0/433 (0) | 1/447 (1)
Upper respiratory tract infection (Infections and infestations) | 0/433 (0) | 2/447 (2)
Urinary tract infection (Infections and infestations) | 3/433 (3) | 3/447 (3)
Wound infection (Infections and infestations) | 1/433 (1) | 0/447 (0)
Chest injury (Injury, poisoning and procedural complications) | 1/433 (2) | 0/447 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Fall (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Lung injury (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Overdose (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Poisoning (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1/433 (1) | 0/447 (0)
Blood bilirubin increased (Investigations) | 1/433 (1) | 0/447 (0)
Blood creatinine increased (Investigations) | 2/433 (2) | 1/447 (1)
Blood urea increased (Investigations) | 1/433 (1) | 0/447 (0)
C-reactive protein increased (Investigations) | 0/433 (0) | 1/447 (1)
Platelet count decreased (Investigations) | 1/433 (1) | 1/447 (1)
Weight decreased (Investigations) | 0/433 (0) | 1/447 (1)
White blood cell count decreased (Investigations) | 0/433 (0) | 1/447 (1)
Anorexia (Metabolism and nutrition disorders) | 2/433 (2) | 0/447 (0)
Dehydration (Metabolism and nutrition disorders) | 6/433 (6) | 4/447 (5)
Fluid retention (Metabolism and nutrition disorders) | 1/433 (1) | 0/447 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2/433 (2) | 0/447 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2/433 (2) | 0/447 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6/433 (6) | 5/447 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/433 (0) | 2/447 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3/433 (3) | 1/447 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/433 (0) | 1/447 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/433 (1) | 0/447 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1/433 (1) | 0/447 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/433 (0) | 1/447 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/433 (1) | 0/447 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/433 (0) | 1/447 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/433 (0) | 1/447 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/433 (1) | 0/447 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/433 (1) | 0/447 (0)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/433 (1) | 0/447 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/433 (1) | 0/447 (0)
Ataxia (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Carotid artery occlusion (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Cerebral haemorrhage (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Convulsion (Nervous system disorders) | 2/433 (2) | 6/447 (6)
Diplegia (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Encephalopathy (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Epilepsy (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Hemiparesis (Nervous system disorders) | 0/433 (0) | 1/447 (1)
Lethargy (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Nervous system disorder (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Speech disorder (Nervous system disorders) | 0/433 (0) | 1/447 (1)
Spinal cord compression (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Transient ischaemic attack (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Unresponsive to stimuli (Nervous system disorders) | 1/433 (1) | 0/447 (0)
Vocal cord paralysis (Nervous system disorders) | 0/433 (0) | 1/447 (1)
Confusional state (Psychiatric disorders) | 1/433 (1) | 2/447 (2)
Insomnia (Psychiatric disorders) | 1/433 (1) | 1/447 (1)
Panic attack (Psychiatric disorders) | 1/433 (1) | 0/447 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 1/433 (1) | 0/447 (0)
Haematuria (Renal and urinary disorders) | 0/433 (0) | 1/447 (1)
Renal failure (Renal and urinary disorders) | 5/433 (5) | 1/447 (1)
Renal failure acute (Renal and urinary disorders) | 2/433 (2) | 1/447 (1)
Urinary retention (Renal and urinary disorders) | 0/433 (0) | 2/447 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 1/447 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15/433 (16) | 15/447 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0/433 (0) | 1/447 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3/433 (3) | 3/447 (3)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0/433 (0) | 1/447 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 3/447 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 0/447 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 1/447 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/433 (0) | 1/447 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 1/447 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/433 (2) | 3/447 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/433 (0) | 2/447 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 1/447 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1/433 (1) | 1/447 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4/433 (4) | 0/447 (0)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0/433 (0) | 1/447 (1)
Hypotension (Vascular disorders) | 0/433 (0) | 1/447 (1)
Pelvic venous thrombosis (Vascular disorders) | 0/433 (0) | 1/447 (1)
Shock haemorrhagic (Vascular disorders) | 0/433 (0) | 1/447 (1)
Superior vena caval occlusion (Vascular disorders) | 4/433 (4) | 2/447 (2)
Thrombophlebitis superficial (Vascular disorders) | 1/433 (1) | 0/447 (0)
Thrombosis (Vascular disorders) | 1/433 (1) | 0/447 (0)
Vascular insufficiency (Vascular disorders) | 1/433 (1) | 0/447 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin | Etoposide + Carboplatin
Anaemia (Blood and lymphatic system disorders) | 135/433 (175) | 155/447 (200)
Leukopenia (Blood and lymphatic system disorders) | 33/433 (67) | 86/447 (179)
Neutropenia (Blood and lymphatic system disorders) | 82/433 (141) | 252/447 (524)
Thrombocytopenia (Blood and lymphatic system disorders) | 61/433 (117) | 94/447 (151)
Coronary artery disease (Cardiac disorders) | 23/433 (23) | 24/447 (24)
Hypothyroidism (Endocrine disorders) | 26/433 (26) | 12/447 (12)
Abdominal pain (Gastrointestinal disorders) | 24/433 (26) | 27/447 (27)
Constipation (Gastrointestinal disorders) | 135/433 (165) | 124/447 (155)
Diarrhoea (Gastrointestinal disorders) | 62/433 (72) | 59/447 (69)
Dyspepsia (Gastrointestinal disorders) | 24/433 (24) | 24/447 (26)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 28/433 (28) | 21/447 (21)
Nausea (Gastrointestinal disorders) | 166/433 (261) | 159/447 (267)
Stomatitis (Gastrointestinal disorders) | 22/433 (23) | 15/447 (19)
Vomiting (Gastrointestinal disorders) | 71/433 (96) | 72/447 (106)
Asthenia (General disorders) | 48/433 (55) | 43/447 (51)
Chest pain (General disorders) | 98/433 (104) | 114/447 (127)
Fatigue (General disorders) | 153/433 (177) | 182/447 (221)
Mucosal inflammation (General disorders) | 22/433 (26) | 26/447 (33)
Oedema peripheral (General disorders) | 38/433 (40) | 33/447 (41)
Pyrexia (General disorders) | 26/433 (29) | 49/447 (59)
Haemoglobin decreased (Investigations) | 22/433 (24) | 15/447 (15)
Weight decreased (Investigations) | 60/433 (64) | 50/447 (53)
Anorexia (Metabolism and nutrition disorders) | 108/433 (130) | 98/447 (120)
Diabetes mellitus (Metabolism and nutrition disorders) | 45/433 (45) | 44/447 (44)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 45/433 (45) | 47/447 (47)
Hyperglycaemia (Metabolism and nutrition disorders) | 23/433 (25) | 18/447 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 23/433 (24) | 17/447 (18)
Hyponatraemia (Metabolism and nutrition disorders) | 25/433 (31) | 27/447 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23/433 (24) | 38/447 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 61/433 (67) | 81/447 (91)
Bone pain (Musculoskeletal and connective tissue disorders) | 15/433 (16) | 26/447 (26)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23/433 (23) | 31/447 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29/433 (30) | 17/447 (18)
Dizziness (Nervous system disorders) | 30/433 (34) | 41/447 (43)
Headache (Nervous system disorders) | 49/433 (62) | 61/447 (78)
Anxiety (Psychiatric disorders) | 45/433 (45) | 36/447 (36)
Depression (Psychiatric disorders) | 41/433 (41) | 38/447 (38)
Insomnia (Psychiatric disorders) | 72/433 (78) | 68/447 (78)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 69/433 (69) | 71/447 (71)
Cough (Respiratory, thoracic and mediastinal disorders) | 210/433 (218) | 221/447 (239)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 49/433 (50) | 42/447 (43)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 178/433 (189) | 182/447 (200)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 33/433 (34) | 32/447 (34)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 31/433 (31) | 20/447 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 27/433 (29) | 156/447 (158)
Rash (Skin and subcutaneous tissue disorders) | 23/433 (24) | 25/447 (36)
Hypertension (Vascular disorders) | 180/433 (181) | 172/447 (175)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days